CLINICAL TRIAL: NCT03815734
Title: Effects of Motor Imagery on Trapeziometacarpal Osteoarthritis in Women During the Postoperative Immobilization Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Prado Robles (Other)
Responsible Party: Sponsor-Investigator, Eva Prado Robles, Principal investigator. Occupational Therapy, Universidad de León
Organization: Universidad de León (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SALUDDOCTORADO
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis Thumb; Immobilization
Keywords: Mental practice; motor imagery; trapeziometacarpal osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Non intervention group
- intervention group (Experimental): motor imagery group
  Interventions: Procedure: motor imagery

INTERVENTIONS:
Procedure: motor imagery — motor imagery during the postoperative immobilization period
  Arms: intervention group

SUMMARY:
The aim of this study is to verify whether after trapeziometacarpal osteoarthrosis surgery and during the period of immobilization immediately after it, applying motor imagery, improvements are achieved on pain, strength, edema and / or inflammation, function and the joint range, accelerating the recovery process.

DETAILED DESCRIPTION:
Motor imagery (IM) consists of a complex cognitive operation by which an action is simulated without doing it physically.

Many studies support the usefulness of motor imaging in rehabilitation after manual surgery.

An approach based on motor imagery may be useful in trapeziometacarpal osteoarthritis, and may be used to promote motor recovery after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participants on the surgical waiting list of the Hospital of León

Exclusion Criteria:

* Other hand pathologies

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change from Preoperative pain to postoperative pain | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  Visual Analogue Scale (VAS). "0" (better) to "10" (worse)

SECONDARY OUTCOMES:
Mobility of hand | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  Kapandji test
Joint mobility | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  Goniometer
Strength | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  Baseline Pinch Gauge, Hydraulic.
Edema/inflammation | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  Measuring tape. Centimeter measurement. Wrist and thumb perimeter
Quality of life and function | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  The Disabilities of the Arm, Shoulder and Hand questionnaire (DASH). 30-item disability/symptom scale, scored 0 (no disability) to 100
Manual function | 2 weeks before the surgery/5, 7 and 11 weeks after surgery
  The Cochin Hand Functional Scale (CHFS) questionnaire. "0" better to "90" worse

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Seco Calvo, Study Director — Universidad de León
Locations (1):
- Eva, León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stenekes MW, Geertzen JH, Nicolai JP, De Jong BM, Mulder T. Effects of motor imagery on hand function during immobilization after flexor tendon repair. Arch Phys Med Rehabil. 2009 Apr;90(4):553-9. doi: 10.1016/j.apmr.2008.10.029. PMID 19345768
- [Derived] Prado-Robles E, Delgado-Gil JA, Navarro-Prada SR, Rodriguez-Martin B, Gomez-Martinez M, Seco-Calvo J. The effects of motor imagery on trapeziometacarpal osteoarthritis in women during the post-surgical immobilisation period: A protocol for a randomised clinical trial. Br J Occup Ther. 2023 Aug;86(8):531-539. doi: 10.1177/03080226221137771. Epub 2022 Dec 29. PMID 40337611